CLINICAL TRIAL: NCT04223115
Title: Randomized Controlled Trial of Digitalized Cognitive Behavioral Therapy With Telephone Coaching for Mothers Suffering From Depression During Pregnancy
Brief Title: A Randomized Controlled Study of Digitalized Cognitive Behavioral Intervention for Antenatal Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Andre Sourander, Professor, Child Psychiatry, University of Turku
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DEPMOM-2020
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Depression; Antenatal Depression
Keywords: digital intervention; cognitive behavioral therapy; antenatal depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digitalized CBT intervention with phone coaching (Experimental): Participants receive weekly sessions of internet-based CBT, including telephone coaching
  Interventions: Behavioral: Digitalized CBT with phone coaching
- Psychoeducation about depression (Active Comparator): Participants receive psychoeducative material about depression in digitalized form.
  Interventions: Other: Psychoeducation about depression

INTERVENTIONS:
Behavioral: Digitalized CBT with phone coaching — Digitally delivered CBT intervention with weekly phone coaching
  Arms: Digitalized CBT intervention with phone coaching
Other: Psychoeducation about depression — Psychoeducational material about depression in a digitalized form
  Arms: Psychoeducation about depression

SUMMARY:
The main objective of the current research project is to evaluate the effectiveness of the digitalized cognitive behavioral therapy program including telephone coaching for antenatal depressive symptoms. The participants are screened from the general population of pregnant women, as a part of the routine maternity health care check-ups. Mothers with depressive symptoms will be randomized into intervention group receiving guided digitalized treatment program or control group receiving education material about depression in digital form.

ELIGIBILITY:
Inclusion Criteria:

* fluent in written and spoken Finnish or Swedish
* access to computer or mobile phone with internet
* between 12 and 22 weeks pregnant
* screening and baseline score on the EPDS ≥10 points

Exclusion Criteria:

* lifetime history of psychotic disorder (e.g. schizophrenia, schizoaffective disorder, bipolar disorder, psychotic depression)
* active suicidal ideation
* severe substance abuse or dependence
* actively ongoing psychotherapy
* participates in another intervention study aiming at treating the symptoms of antenatal depression
* multiple pregnancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 634 (Estimated)
Dates: Start 2021-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in the Edinburgh Postnatal Depression Scale (EPDS) | Baseline and 11 weeks after randomization
  EPDS is a ten-item self-report questionnaire originally developed to screen for postpartum depression. The respondents are asked about the symptoms of depression. The total score ranges from 0 to 30.

SECONDARY OUTCOMES:
Change in the General Anxiety Disorder 7-item scale (GAD-7) | Baseline and 11 weeks after randomization
  To assess the change in anxiety symptoms from baseline to follow-up, we will use the Generalized Anxiety Disorder 7-item Scale (GAD-7) (Spitzer, Kroenke, Williams, & Löwe, 2006), which is a brief screening measure including seven items asking about anxiety symptoms experienced in the previous two weeks.
Change in the Beck Depression Inventory II (BDI-II) | Baseline and 11 weeks after randomization
  To assess the change in depressive symptoms BDI-II will be used.
Social Phobia Inventory (SPIN) | Baseline and 11 weeks after randomization
  To assess the change in Social Phobia SPIN will be used
Pregnancy-Related Anxiety Questionnaire-Revised (PRAQ) | Baseline and 11 weeks after randomization
  To assess the change in pregnancy related anxiety PRAQ will be used
Perceived Stress Scale (PSS) | Baseline and 11 weeks after randomization
  To assess the change in perceived stress PSS will be used

CONTACTS AND LOCATIONS:
Overall Officials: Andre Sourander, Professor, Principal Investigator — University of Turku, Research Center for Child Psychiatry
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sourander A, Korpilahti-Leino T, Ristkari T, Koffert T, Arrhenius B, Stahlberg T, Hinkka-Yli-Salomaki S, Berglund M, Upadhyaya S, Wan Mohd Yunus WMA, Sinokki A, Hagg R, Marjamaki A, Kankaanranta I, Palmroth J, Sourander S, Zadkova A, Casagrande L, Yamada Y, Karjalainen S, Matinolli HM, Vuori M. Internet-assisted cognitive behavioral therapy with telephone coaching versus an educational control for antenatal depression: protocol for a randomized controlled trial with population-based screening. Front Psychiatry. 2025 Nov 3;16:1604352. doi: 10.3389/fpsyt.2025.1604352. eCollection 2025. PMID 41256941